CLINICAL TRIAL: NCT07130851
Title: Mapping of Vestibular Center Activation Using fMRI in Patients With Vestibular Schwannoma
Brief Title: Mapping of Vestibular Centers Activation Using fMRI in Patients With Vestibular Schwannoma
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Marketa Bonaventurova (Other)
Responsible Party: Sponsor-Investigator, Marketa Bonaventurova, MD, Charles University, Czech Republic
Organization: Charles University, Czech Republic (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EK-279.4/24
Record Dates: First submitted 2025-07-05; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Vestibular Schwannoma; Unilateral Vestibular Deficit; Healthy
Keywords: vestibular centers; functional magnetic resonance; vestibular schwannoma; central compensation
MeSH Terms: conditions — Neuroma, Acoustic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vetibular schwannoma patients (Experimental): Patients with vestibular schwannoma undergoing surgical removal of the tumor one day before the surgery: objective methods videoHead Impulse test, cervical vestibular evoked myogenic potentials, air calorics, clinical otoneurologic examination, functional magnetic resonance subjective methods: questionnaires (DHI,..) one week after the surgery: objective methods videoHead Impulse test, clinical otoneurologic examination, functional magnetic resonance subjective methods: questionnaires (DHI,..)
  Interventions: Procedure: vestibular schwannoma resection
- Healthy controls (No Intervention): The healty patients without the history of vestibular disorder. objective methods videoHead Impulse test, cervical vestibular evoked myogenic potentials, functional magnetic resonance subjective methods: questionnaires (DHI,..)

INTERVENTIONS:
Procedure: vestibular schwannoma resection — Vestibular schwannoma resection leads to partial or combined acute unilateral peripheral or combined vestibular lesion.The organism responds with the process of central vestibular compensation.
  Arms: Vetibular schwannoma patients

SUMMARY:
The goal of this clinical trial is to visualize the possible activation of vestibular centers in the brain using in patiens with unilateral vestibular damage, specifically in patients after vestibular schwannoma surgery.

The main questions it aims to answer are:

1. Is there a difference in the proces sof activation of vestibular centers in patients with unilateral vestibular disorder and healthy subjects.
2. Are we able to effect this activation with our postoperative treatment? Researchers will compare the obtained results between patients with unilateral vestibular disorder and healthy controls.

Participants will be asked to fill out the set of questionaires, to undergo clinical objective vestibular examnation and examination in magnetic resonance.

ELIGIBILITY:
Inclusion Criteria:

* vestibular schwannoma

Exclusion Criteria:

* claustrophobia, visual impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Identification of cortical vestibular center in acute unilateral vestibular lesion | baseline and one week
  Fuctional magnetic resonance (fMRI) could display certain areas of the brain and its pathways involved in the process of central compensation resulting from the acute unilateral vestibular lesion.
  We aim to compare pre- and post- operative fMRI results with the results of healthy controls to see whether there is a difference in activating vestibular centers and maintaining the equilibrium after the central compensation occurs. Different level of activation of vestibular cortical areas, resp. differences in activation in response to optokinetic stimulation will be measured in healthy controls and study group. Evaluation of functional brain MRI will be provided by expert neuroradiologist. Vestibular function will be assessed by objective vestibular tests (videonystagmography, video Head Impuls Test) and by subjective scales (questionnaires - The Penn Acoustic Neuroma Quality-of-Life scale, Dizziness Handicap Inventory - in both the higher score indicates higher handicap).

SECONDARY OUTCOMES:
Change in cortical activation in response to acute onset of vestibular loss | baseline and one week
  Evaluation of differences between control and study group in functional brain MRI in response to wide field optokinetic stimulation. Differences in size and level of activation of vestibular cortical areas will be evaluated by expert neuroradiologist.
Possible influence of vestibular training in virtual reality environment on the rate of vestibular center activation | baseline and 3 months
  The cohort group, which undergoes vestibular rehabilitation in virtual reality environment, will be evaluated and compared to control and study group. Functional brain MRI in response to wide field optokinetic stimulation will be evaluated by expert neuroradiologist.
  The obtained data could serve as a basis for understanding the possibility of influencing the central compensation process and potentially, in the future, utilizing virtual reality as a tool for vestibular training.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Otorhinolaryngology and Head and Neck Surgery, 1st Medical Faculty Charles University and University Hospital Motol, Prague, Czechia

IPD SHARING:
Plan to Share IPD: Yes
IPD used in the results publication
Supporting Information: Study Protocol

REFERENCES:
- [Background] Hufner K, Stephan T, Hamilton DA, Kalla R, Glasauer S, Strupp M, Brandt T. Gray-matter atrophy after chronic complete unilateral vestibular deafferentation. Ann N Y Acad Sci. 2009 May;1164:383-5. doi: 10.1111/j.1749-6632.2008.03719.x. PMID 19645932
- [Background] Helmchen C, Klinkenstein JC, Kruger A, Gliemroth J, Mohr C, Sander T. Structural brain changes following peripheral vestibulo-cochlear lesion may indicate multisensory compensation. J Neurol Neurosurg Psychiatry. 2011 Mar;82(3):309-16. doi: 10.1136/jnnp.2010.204925. Epub 2010 Aug 27. PMID 20802221